CLINICAL TRIAL: NCT04208373
Title: A Phase 1, Open-label, Fixed-sequence, 2-Panel Study to Assess the Effects of Itraconazole and Etravirine on the Single-dose Pharmacokinetics of JNJ-64417184 in Healthy Adult Subjects
Brief Title: A Study to Assess the Effects of Itraconazole and Etravirine on JNJ-64417184 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108747; 2019-003928-20 (EudraCT Number); 64417184RSV1002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-12-20; First posted 2019-12-23 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — Itraconazole; etravirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Panel 1: JNJ 64417184 plus Itraconazole (Experimental): Participants will receive single oral dose of JNJ 64417184 on Day 1 followed by itraconazole once daily on Days 6 to 13 along with a single dose of JNJ 64417184 on Day 9 orally.
  Interventions: Drug: JNJ-64417184; Drug: Itraconazole
- Panel 2: JNJ 64417184 plus Etravirine (Experimental): Participants will receive single oral dose of JNJ-64417184 on Day 1 followed by etravirine twice daily on Days 6 to 19 along with single dose of JNJ 64417184 on Day 15.
  Interventions: Drug: JNJ-64417184; Drug: Etravirine

INTERVENTIONS:
Drug: JNJ-64417184 — JNJ 64417184 tablets will be administered orally.
Drug: Itraconazole — Itraconazole capsules will be administered orally
  Arms: Panel 1: JNJ 64417184 plus Itraconazole
Drug: Etravirine — etravirine tables will be administered orally.
  Arms: Panel 2: JNJ 64417184 plus Etravirine

SUMMARY:
The main purpose of this study is to evaluate the effects of itraconazole or etravirine on the single-dose pharmacokinetics (PK) of JNJ 64417184 in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (weight [kg]/height2 [m]2) between 18.0 and 30.0 kg/m2, extremes included, and body weight not less than 50 kg at screening
* Healthy on the basis of physical examination, medical and surgical history, and vital signs (systolic blood pressure, diastolic blood pressure, and pulse rate [after the participant is supine for at least 5 minutes], respiratory rate, and oral body temperature) performed at screening. If there are abnormalities, the participant may be included only if the investigator judges the abnormalities to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* Female participant must have a negative highly sensitive serum beta human chorionic gonadotropin pregnancy test at screening and a negative urine pregnancy test on Day 1
* Female participant must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for at least 90 days after the last study drug intake
* Must not use nicotine-containing substances including tobacco products (example, cigarettes, e-cigarettes, cigars, chewing tobacco, gum, or patch) for at least 3 months prior to screening

Exclusion Criteria:

* History of liver or renal dysfunction (calculated creatinine clearance/estimated glomerular filtration rate (eGFR) less than (<) 60 milliliter per minute (mL/min) at screening, calculated by the Modification of Diet in Renal Disease [MDRD] formula), significant cardiac, vascular, pulmonary, gastrointestinal (such as significant diarrhea, gastric stasis, or constipation that in the investigator's opinion could influence drug absorption or bioavailability), endocrine, neurologic, hematologic, rheumatologic, psychiatric, neoplastic, or metabolic disturbances
* - Past history of cardiac arrhythmias (example, extrasystoli, tachycardia at rest), history of risk factors for Torsade de Pointes syndrome (example, hypokalemia, family history of long QT Syndrome)
* Any evidence of heart block or bundle branch block at screening
* Current human immunodeficiency virus (HIV)-1 or HIV-2 infection (confirmed by antibodies) at screening
* History of hepatitis A virus immunoglobulin M antibody, hepatitis B surface antigen, or hepatitis C virus antibody positive, or other clinically active liver disease, or tests positive for hepatitis A virus immunoglobulin M antibody, hepatitis B surface antigen, or hepatitis C virus antibody at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Analyte concentration (Cmax) of JNJ 64417184 | Predose up to 144 hours post dose
  Cmax is defined as maximum observed plasma analyte.
Area Under the Concentration-time Curve from Time Zero to the Last Measurable Concentration (AUC [0-last]) of JNJ 64417184 | Predose up to 144 hours post dose
  AUC (0-last) is defined as the area under the plasma analyte concentration- time curve (AUC) from time 0 to the time of the last measurable (non-below qualification limit) concentration.
Area Under the Concentration-time Curve from Time Zero to Infinity (AUC [0-infinity]) of JNJ 64417184 | Predose up to 144 hours post dose
  AUC (0-infinity) is defined as AUC from time 0 to infinite time, calculated as the sum of AUC(0-last) and C(last)/ lambda(z), wherein C(last) is the last observed quantifiable concentration; extrapolations of more than 20 percent (%) of the total AUC.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AE) as a Measure of Safety and Tolerability | Up to 54 days
  An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- SGS Clinical Pharmacology Unit (located in ZNA Stuivenberg), Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency